CLINICAL TRIAL: NCT06709703
Title: L'Alignement cinématique Dans Les prothèses de Totales de Genou : un Essai randomisé contrôlé à Double Insu Comparant la Robotique Aux Instruments Traditionnels
Brief Title: Kinematic Alignment in Total Knee Arthroplasty - a Double-blind Randomised Controlled Trial Between Robotic and Caliper-based Techniques
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Hopital Charles Lemoyne (Other)
Responsible Party: Principal Investigator, Samuel Larrivée, Orthopaedic Surgeon, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-958
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Arthritis; Arthritis (Knee); Osteoarthritis; Osteoarthritis Knee Pain; OA; OA Knee; OA Knee Pain; Osteoarthritis of Knee; Gonarthrosis; Primary
Keywords: osteoarthritis; arthritis; knee osteoarthritis; knee OA; knee arthritis; total knee replacement; robotic; kinematic alignment; patient-specific surgery
MeSH Terms: conditions — Arthritis; Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled-trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician will be blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Kinematic knee replacement with traditional instruments (Active Comparator): Patients will undergo kinematic aligned knee replacement done using traditional instruments and cut guides
  Interventions: Procedure: Kinematic aligned total knee replacement
- Robotic-assisted kinematic knee replacement (Experimental): Patients will undergo kinematic aligned knee replacement done using robotic assistance
  Interventions: Procedure: Kinematic aligned total knee replacement

INTERVENTIONS:
Procedure: Kinematic aligned total knee replacement — Replacement of worn knee cartilage using a prosthesis. The alignment is determined according to the patient's anatomy and ligament balance.

SUMMARY:
Knee replacement surgery is a surgery designed to treat severe arthritis of the knee. However, as many as 20% of patients are not satisfied with the results of their surgery. To place the knee replacement in correct position, the kinematic alignment method, which tries to reproduce the patient normal anatomy, has shown promise in improving the satisfaction after knee replacement surgery. It is not known if using a robotic arm to assist in surgery is better than the traditional method when trying to recreate kinematic alignment.

The goal of this study is to learn if robotic assisted surgery is better than traditional method for knee replacement done using kinematic alignment. The main questions the study tries to answer are:

1. Do the radiographs of kinematic knee replacement surgeries done with robotic assistance show better alignment than radiographs of kinematic knee replacements done with the traditional method?
2. Does robotic assisted kinematic knee replacement give better function to patients than traditional knee replacement done with kinematic alignment?
3. Does robotic assisted kinematic knee replacement decrease pain, improve knee movement and improve knee stability better than traditional knee replacement done with kinematic alignment?
4. Are there more complications with robotic assisted kinematic knee replacement in comparison to traditional kinematic knee replacement?
5. How long long does it take a surgeon to become good a performing a kinematic knee replacement using robotic assistance? Researchers will compare knee replacements done using a robotic to make the bone cuts, and compare it to the usual method using guides and manual instruments. All the knee replacements will be done using the kinematic alignment and with the same type of knee replacement prothesis.

Participants will:

* Have a knee replacement done with the kinematic alignment technique by an experienced surgeon, with or without robotic assistance during the surgery.
* Visit the clinic before surgery, six weeks after surgery, three months, six months, twelve months and twenty-four months after the surgery.
* Fill questionnaire, have their knee examined and have radiographs of their knee done at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or above
* Patient being consented for a primary total knee arthroplasty (TKA)
* The primary TKA is planned to be done with kinematic alignment
* All pre-operative alignments are included

Exclusion Criteria:

* Revision TKA (including revision of unicompartimental knee arthroplasty into total knee arthroplasty with primary components). TKA being done in the setting of previous femur or tibia fracture or osteotomy are however included.
* No available adequate pre-operative imaging
* Patient who does want to be randomized of the two groups
* At the discretion of the surgeon, if the patient's pathology or particular anatomy precludes the use of kinematic alignment technique, robotic surgery, or traditional instrument TKA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Radiographic alignment of the knee | Pre-operative alignement and 6 months post-operative alignement.
  Long leg anteroposterior views of both legs and lateral knee radiographs will be used to measure knee alignment and position of the knee replacement hardware. The angles measured and analyzed will be:
  * The hip-knee-ankle (HKA) angle
  * Medial proximal tibia mechanical angle (MPTAm)
  * Lateral distal femur mechanical angle (LDTAm)
  * Distal femur flexion angle (DFFA)
  * Posterior tibial slope (PTS) Radiographic measurements will be made by a trained observer and a fellowship-train arthroplasty surgeon.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-operative, 6 weeks, 6 months, 12 months, 24 months post-operative
  Patient questionnaire (42 questions) evaluating knee pain, symptoms, function, recreational activities and knee-related quality of life. The questionnaire is score over 100 points, with a higher score meaning better knee function.
Forgotten joint score | Pre-operative, 6 weeks, 6 months, 12 months and 24 months post-op
  A 12-questions form asking patients if they forget about their joint during activities of daily living.
Joint perception question | Pre-operative, 6 weeks, 6 months, 12 months and 24 months post-operative
  A single item question asking participants how they perceive their operated knee, from "like a native or natural joint" to "like a nonfunctional joint".

SECONDARY OUTCOMES:
Pain visual analog scale | Pre-op, 6 weeks, 6, 12, 24 months
  Pain rated on a 10 cm visual analog scale from "no pain" to "worst pain imaginable"
Subjective Assessment Numeric Evaluation Scale (SANE) | Pre-op, 6 weeks, 6, 12, 24 months
  Single question evaluation scale asking the patient to rate their knee function from 0 (no function) to 100 (completely normal function)
Knee range of motion | Pre, 6 weeks, 6 and 12 months post-op
  Maximum passive flexion and extension measured with goniometer
Knee stability | Pre-op, 6 weeks, 6 and 12 months post-op
  Anterior drawer, posterior drawer, valgus stress, varus stress. Instability rated for each test 1 to 3 by treating surgeon.

OTHER OUTCOMES:
Intra-operative procedures | At the time of surgery
  During surgery, the knee for additional intra-operative procedures to obtain a stable knee replacement will be noted:
  * Need for ligamentous release - lateral release, medial release, lateral retinaculum release, posterior cruciate ligament release
  * Need for tibial or femoral recut
Surgical cost | At the time of surgery
  Total cost of implants and equipment used will be calculated at the end of each surgical case.
Surgical time | At the time of surgery
  The time from first incision to skin closure will be noted at each surgery.
Intra-operative complications | At the time of surgery
  The incidence of intra-operative complications will be noted:
  * Unplanned ligament injury
  * Neurovascular damage
  * Intra-operative tibial of femoral fracture
  * Any other complications noted during surgery

IPD SHARING:
Plan to Share IPD: No
Anonymous individual patient data will be shared only with a direct request to the study principal investigator.

REFERENCES:
- [Background] Zhang J, Ndou WS, Ng N, Gaston P, Simpson PM, Macpherson GJ, Patton JT, Clement ND. Robotic-arm assisted total knee arthroplasty is associated with improved accuracy and patient reported outcomes: a systematic review and meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2022 Aug;30(8):2677-2695. doi: 10.1007/s00167-021-06464-4. Epub 2021 Feb 6. PMID 33547914
- [Background] Agarwal N, To K, McDonnell S, Khan W. Clinical and Radiological Outcomes in Robotic-Assisted Total Knee Arthroplasty: A Systematic Review and Meta-Analysis. J Arthroplasty. 2020 Nov;35(11):3393-3409.e2. doi: 10.1016/j.arth.2020.03.005. Epub 2020 Mar 11. PMID 32234326
- [Background] Van Essen J, Stevens J, Dowsey MM, Choong PF, Babazadeh S. Kinematic alignment results in clinically similar outcomes to mechanical alignment: Systematic review and meta-analysis. Knee. 2023 Jan;40:24-41. doi: 10.1016/j.knee.2022.11.001. Epub 2022 Nov 17. PMID 36403396
- [Background] Dossett HG, Estrada NA, Swartz GJ, LeFevre GW, Kwasman BG. A randomised controlled trial of kinematically and mechanically aligned total knee replacements: two-year clinical results. Bone Joint J. 2014 Jul;96-B(7):907-13. doi: 10.1302/0301-620X.96B7.32812. PMID 24986944
- [Background] Turan K, Camurcu Y, Kezer M, Uysal Y, Kizilay YO, Ucpunar H, Temiz A. A comparison of robotic-assisted and manual techniques in restricted kinematically aligned total knee arthroplasty: coronal alignment improvement with no significant clinical differences. Knee Surg Sports Traumatol Arthrosc. 2023 Nov;31(11):4673-4679. doi: 10.1007/s00167-023-07426-8. Epub 2023 May 10. PMID 37165209